CLINICAL TRIAL: NCT03697720
Title: Examining the Role of Improved NSAID Management in Treating Dysmenorrhea and Bladder Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Frank Tu, Division Director MIS/Clinical Professor, Endeavor Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EH18-128
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-09

CONDITIONS: Dysmenorrhea; Pain
Keywords: cross-organ sensitivity; bladder pain; NSAID; visceral pain
MeSH Terms: conditions — Dysmenorrhea; Pain; Visceral Pain | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Primary Dysmenorrhea (Experimental): We will look at the effects of naproxen 500mg use on pain starting just before and during menses.
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Naproxen — Participants will take naproxen 500mg BID before and for the first 3 days of their period.

SUMMARY:
The goal of this study is to see if optimized use of naproxen for treatment of dysmenorrhea will improve pain report from baseline. In addition, we will determine whether cross-organ influences from the uterus on bladder pain sensitivity change from baseline after reduced menstrual pain experience over six months. Finally, a battery of quantitative sensory tests and EEG measures of sensory sensitivity will be used to evaluate mechanisms associated with improvements in menstrual and bladder pain.

DETAILED DESCRIPTION:
Endometrial shedding during the menstrual cycle elicits profound changes in neuronal activity and cytokine concentrations producing moderate to severe pelvic pain in more than 20% of reproductive-age women. One out of every five of those women in turn will experience chronic pelvic pain (CPP) which may be in part due to cross-organ neural sensitization.

In this study we will establish whether prophylactic and adequate dosages of naproxen are capable of reducing menstrual pain more than *** use.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive-age women (age 18-45) with dysmenorrhea
* Average menstrual pain ≥ 5/10 (0=no pain and 10=the worst imaginable pain) on at least one day during menses or during withdrawal uterine bleeding from cyclic OCs without painkillers
* Menstrual pain in the region between the umbilicus and the perineum, above the level of the inguinal ligament
* Indication the participant has attempted to resolve pain by medical means (including NSAIDs and/or OCPs)

Exclusion Criteria:

* Presence of active pelvic or abdominal malignancies (primary or metastatic)
* Absence of regular menses (including current pregnancy, recent pregnancy, or active breast feeding)
* Active genitourinary infection in the last four weeks
* Unable to read or comprehend the informed consent in English
* Unwilling to complete study procedures
* Presence of hypertension or risk for developing hypertension
* Unwillingness to take naproxen and/or placebo
* Contradictions to taking naproxen (allergies, kidney disease, anemia, alcoholism, cardiovascular disease, stomach or intestinal ulcer or abnormal liver function)
* Formal urological diagnosis such as overactive bladder or bladder pain syndrome.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Tu, MD, MPH, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University Health System, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan WY, Dawood MY, Fuchs F. Prostaglandins in primary dysmenorrhea. Comparison of prophylactic and nonprophylactic treatment with ibuprofen and use of oral contraceptives. Am J Med. 1981 Mar;70(3):535-41. doi: 10.1016/0002-9343(81)90576-3. PMID 7011011
- [Background] Oladosu FA, Tu FF, Hellman KM. Nonsteroidal antiinflammatory drug resistance in dysmenorrhea: epidemiology, causes, and treatment. Am J Obstet Gynecol. 2018 Apr;218(4):390-400. doi: 10.1016/j.ajog.2017.08.108. Epub 2017 Sep 6. PMID 28888592
- [Background] Tu FF, Datta A, Atashroo D, Senapati S, Roth G, Clauw DJ, Hellman KM. Clinical profile of comorbid dysmenorrhea and bladder sensitivity: a cross-sectional analysis. Am J Obstet Gynecol. 2020 Jun;222(6):594.e1-594.e11. doi: 10.1016/j.ajog.2019.12.010. Epub 2019 Dec 20. PMID 31870730

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between April 2018 and December 2019 from our registry and other studies.
Period: Overall Study
Arm/Group | Primary Dysmenorrhea
Started | 26
Completed | 19
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Primary Dysmenorrhea
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 17
  More than one race | 2
  Unknown or Not Reported | 0
Menstrual Pain [Mean (Standard Deviation); unit: Numerical rating scale] — Numeric Rating Scale is a 0-10 scale with 0 being no pain and 10 being the worst imaginable. Results from the NRS for worst day's menstrual pain are reported
  Numerical rating scale | 6.0 (2.0)
Bladder Pain [Mean (Standard Deviation); unit: Visual Analog Scale 0-100] — Visual analog scale is a 0-100 scale with 0 being no pain and 100 worst pain imaginable. Results from the VAS of the bladder filling test are compared to determine if participants had a reduction in pain following treatment. Bladder pain ratings at first urge are used as the outcome measure. Population: 3 participants did not complete baseline visits to measure bladder pain
  Visual Analog Scale 0-100
    number analyzed (Participants) | 23
    (all) | 16.5 (16.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Menstrual Pain
Description: Score on a scale. Specifically, we used a Numeric Rating Scale (NRS)- 0 through 10 scale with 0 being no pain and 10 worst pain imaginable. Results for the worst menstrual pain score on an NRS from the 6-8 mth menstrual pain diary will be compared to baseline pretreatment diary worst pain score.
Time Frame: 6-8 months
Population: Some participant data were missing due to attrition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Dysmenorrhea
Number analyzed (Participants) | 19
score on a scale | 4.1 (2.4)
Statistical Analysis 1: Comparison: Primary Dysmenorrhea; Paired t-tests were used to compare worst menstrual pain rating across diary day (0-10 numeric rating scale) from baseline and at 6-8 maths followup; Test type: Superiority; p < 0.0001, t-test, 2 sided — The a priori threshold for statistical significance was .05; Paired t-test

2. Primary Outcome: Change in Participant Bladder Pain Sensitivity From Baseline
Description: Score on a scale. Specifically, we used a Visual Analog Scale- 0 through 100 scale with 0 being no pain and 100 worst pain imaginable. Results from the visual analog scale (VAS) of the bladder filling test at the baseline and 6-8 mph followup visit will be compared to determine if naproxen treatment of menstrual pain affected bladder pain. Bladder pain ratings at first urge will be used at the outcome measure.
Time Frame: 6-8 months
Population: Some participant data were missing due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Primary Dysmenorrhea
Number analyzed (Participants) | 17
score on a scale | 10.7 (10.6)
Statistical Analysis 1: Comparison: Primary Dysmenorrhea; Test type: Superiority; p = .119, t-test, 2 sided; paired t-test

ADVERSE EVENTS:
Time Frame: 6 months
Description: Participants were asked to verbally relay any AEs they had experienced during the trial at follow-up. Please note, all-cause mortality or serious & other AEs were not formally queried, but we did monitor for them.
Arm/Group | Primary Dysmenorrhea
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Dysmenorrhea (N=26)
Dyspepsia grade 1 (Gastrointestinal disorders) | 1 (1) — Nausea, upset stomach (mild, grade 1). Mild symptoms; intervention not indicated. Maybe unrelated to study drug as another new drug was being started at the same time.

LIMITATIONS AND CAVEATS:
There was some loss to follow-up. We did not systematically query for adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT03697720/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT03697720/ICF_001.pdf